CLINICAL TRIAL: NCT06529861
Title: Identification of Mechanisms Behind Microvascular Dysfunction in Ischemia With No Obstructive Coronary Artery Disease
Brief Title: Mechanisms Behind Microvascular Dysfunction in INOCA
Acronym: ExINOCA-P1
Status: Not yet recruiting | Type: Observational
Sponsor: Bispebjerg Hospital (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Eva Prescott, MD Clinical Professor, Bispebjerg Hospital
Other Study IDs: ExINOCA - Part I
Record Dates: First submitted 2024-07-08; First posted 2024-07-31 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Coronary Microvascular Dysfunction; Ischaemia With Non Obstructed Coronary Arteries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood sample for biobank: A blood sample will be collected for inclusion in a biobank for future research. As part of this process, a distinct patient information and consent form will be administered.
  Adipose biopsies are assessed in a laboratory at the Biomedical Institute, University of Copenhagen.
  From these biopsies, segments of small arteries will be promptly dissected free. One segment will be mounted in a myograph for recording of isometric tension (i.e., vasoconstriction and vasodilation) and for histochemical analysis, while the other segment will be snap-frozen for proteomic and histological analysis and the adipose tis-sue/perivascular adipose tissue will be used for genomic and transcriptomic analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Ischemia and no obstructive coronary arteries: patients with angina and reduced myocardial blood flow reserve
  Interventions: Diagnostic Test: [15O]H2O-PET Imaging
- Control: controls without angina
  Interventions: Diagnostic Test: [15O]H2O-PET Imaging

INTERVENTIONS:
Diagnostic Test: [15O]H2O-PET Imaging — This imaging technique will be used to measure myocardial blood flow (MBF) and myocardial blood flow reserve (MBFR) in patients. The PET-CT scan involves the use of the radioactive tracer [15O]H2O to visualize blood flow in the heart, providing crucial data on coronary microvascular function.

SUMMARY:
The purpose of the study is to identify the causes of chest pain in patients experiencing chest pain with no signs of narrowing in the coronary arteries of the heart.

DETAILED DESCRIPTION:
A significant number of patients with ischemic heart disease do not exhibit coronary obstruction, leading to their symptoms being attributed to coronary microvascular dysfunction, a condition known as ischemia with no obstructive coronary artery disease (INOCA). Despite a considerable patient population affected by INOCA, the specific mechanisms underlying this microvascular dysfunction are not fully understood, often resulting in a lack of targeted treatment. There is evidence to suggest that exercise capacity is linked to coronary microvascular function, an area yet to be explored.

This study aims to identify mechanisms underlying Coronary microvascular dysfunction (CMD) in angina and to assess whether exercise training can improve the condition. In study part I 30 patients with impaired coronary microvascular function and 30 asymptomatic controls will be studied to identify vascular and related molecular mechanisms underlying INOCA by investigating microvascular function in the heart and in cutaneous tissue, skeletal muscle, and adipose tissue.

ELIGIBILITY:
Inclusion Criteria:

Only for angina patients: Have CMD, defined as myocardial bloodflow re-serve (MBFR) < 2.5 or hyperemic myocardial blood flow (hMBF) < 2.3ml/g/min

Exclusion Criteria:

* Females of childbearing potential (defined as a premeno-pausal female capable of becoming pregnant). The female patient must either be postmenopausal, defined as amen-orrhea for at least 1 year, or surgically sterile
* Heart failure, defined as left ventricular ejection fraction of less than 40%
* Uncontrolled hypertension defined as blood pressure above target 140/90 for all
* Co-morbidity resulting in <1 year expected survival
* Considered by the investigator, for any reason, to be an unsuitable candidate for the study.
* Unable or unwilling to exercise, e.g. due to arthritis or injury*
* Already are regularly physically active and/or have a maximal oxygen uptake >45 ml/kg/min
* The subject has a known allergy to either: norepinephrine, adenosine, ketorolac, and or ascorbic acid (vitamin C).

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Ischemia with no obstruction of coronary arteries (INOCA) is estimated to affect >150.000 Danes and the majority are females. These patients have a shorter life expectancy than age matched controls and a higher incidence of major cardiovascular events (1,2).
  INOCA is caused by microvascular dysfunction. When there is dysfunction in the microvascu-lature, the blood flow within the coronary vessels fails to increase adequately to meet the de-mand, resulting in ischemia and pain (angina).
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2027-10-30 (Estimated); Study Completion 2028-05-15 (Estimated)

PRIMARY OUTCOMES:
Vascular function in response to acetylcholine stress | Baseline only
  Vascular conductance measured by ultrasound doppler during infusion of acetylcholine

SECONDARY OUTCOMES:
Vascular function in response to acetylcholine adenosine stress | Baseline only
  Vascular conductance measured by ultrasound doppler during infusion of Adenosine
Myocardial Blood flow reserve | Baseline only
  Determined by the clinical assessment of [15O]H2O-PET
Skeletal Muscle Microvascular Function | Baseline only
  Evaluated by brachial artery ultrasound Doppler in response to exercise stress to measure blood flow responsiveness in skeletal muscles.
Changes in isolated small artery reactivity assessed with myography | Baseline only
  Analyzed using myograph to study the tone of smooth muscle cells
Arterial Compliance | Baseline only
  Determined by calculations made from intra-arterial pressure and arterial diameter measurements obtained via ultrasound Doppler to assess arterial compliance.
Plasma Lipids | Baseline only
  Conducted through clinical chemical analysis to measure levels of HDL, and triglycerides in the blood, providing insights into lipid profiles.
Plasma HbA1c | Baseline only
  Conducted through clinical chemical analysis to measure levels of HbA1c in the blood, providing insights into glucose metabolism.
Plasma Levels of Markers Related to Vascular Function | Baseline only
  Assessed using Mesoscale/ELISA to quantify biomarkers associated with vascular function
Plasma Levels of Inflammatory Markers | Baseline only
  Measured using Mesoscale/ELISA/O-Link platforms to evaluate the presence and levels of inflammatory markers
Arterial Blood Pressure | Baseline only
  Monitored with automated blood pressure measurements at rest and during exercise to assess overall cardiovascular health and response to physical activity.
Cardiac Function | Baseline only
  Changes in stroke volume using echocardiography during rest and exercise stress

OTHER OUTCOMES:
Tone of smooth muscle cells | Baseline only
  Changes in isolated small artery reactivity assessed with myography
Proteomic and transcriptomic analyses | Baseline only
  Changes in gene and protein expressions patterns in small arteries

CONTACTS AND LOCATIONS:
Overall Officials: Ylva Hellsten, Professor, Study Chair — University of Copenhagen
Locations (1):
- Frederiksberg Hospital, Dept. of Cardiology, Building 16, Y3, Nordre Fasanvej 57, Frederiksberg, Denmark, 2000, Copenhagen, Denmark

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-07-29): https://cdn.clinicaltrials.gov/large-docs/61/NCT06529861/Prot_SAP_000.pdf